CLINICAL TRIAL: NCT02007109
Title: Use of Baxter Animated Retching Faces (BARF) Scale to Measure Nausea in Children Who Speak Spanish
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Mary Felberg, MD, Baylor College of Medicine
Other Study IDs: H32424
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Results first posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nausea measurement by VAS and BARF: All patients will be asked to rate their nausea on both the VAS and the BARF scales. For the nausea scales, the script would be: "Have you thrown up or felt like you were going to throw up before? How did your tummy feel then? We call that feeling of being sick to the stomach as nausea.
  For the BARF scale:These faces show children who feel no nausea at all, who feel a little bit nauseated, who feel even more nauseated, and these are children who have the most nausea it is possible to feel." (Point to the each face at the appropriate time). Which face is more like you feel right now?" For the VAS scale: On this line the far left indicates "No nausea" and the far right" Worst nausea ever." Can you show me on this line how much nausea you have right now?

SUMMARY:
Pediatric research in the management of nausea has been limited by the absence of a reliable method to quantify the intensity of this subjective symptom. In adults, the visual analog scale (VAS) is an accurate tool, but this has not been shown to be reliable in young children. A scale is a series of points made on a line that will be used for measurement; a mark on the far left of the line shows little pain and the mark on the far right means alot of pain.

DETAILED DESCRIPTION:
By default the most common objective outcome measure used in pediatric studies has been the incidence and number of emetic episodes. This measure, however, correlates poorly with the somatic subjective symptom of nausea. Apfel et al have shown that 30-40% of adult patients undergoing surgery have post discharge nausea and / or vomiting while 12% have vomiting. These data on nausea in adults were based on a visual analog scale for nausea. There are no data on the incidence of postoperative nausea in children since the severity of symptoms are difficult to measure as younger children are known to be unable to use the VAS reliably. Recently a pictorial scale for measuring nausea, the Baxter Animated Retching Faces (BARF) scale, has been developed and shown to have construct, content and convergent validity as an instrument to measure nausea in children. This was a two center study that was limited to children who could speak English. The clinical usefulness of this scale in determining the incidence of postoperative and post-discharge nausea in children has yet to be determined including the lowest age where it can be used reliably, the score associated with a patient's perception of a need for treatment, the minimum change in the scores of clinical relevance and the test-retest reliability when nausea is rated as not having changed. The score has also not been validated in children who speak Spanish. This study is designed to provide the missing information and will specifically look at the Spanish speaking population.

ELIGIBILITY:
Inclusion Criteria:

* (1) Spanish speaking children (2) Age > 7 years but below 18 years (3) Elective surgery (4) American Society of Anesthesiologists physical status 1-3 (Free from major concurrent disorders) (5) Free from nausea and / or vomiting in the previous 24 hours (6) Cognitive and communicative ability to rate the intensity of symptoms as described below.

Exclusion Criteria:

* (1) Inability to understand or speak Spanish (2) Developmental delay (3) Blindness (4) Impaired cognitive or communicative abilities including inability to rate the intensity of symptoms (5) Surgical procedure where vision or hearing is anticipated to be impaired in the immediate postoperative period (6) Nausea and /or vomiting within 24 hours of procedure, (7) Patient or parental refusal to participate (8) Pregnant females

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Spanish Speaking patients undergoing surgery
Sampling Method: Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2014-01; Primary Completion 2018-03-08 (Actual); Study Completion 2018-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary A Felberg, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children't Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Watcha MF, Medellin E, Lee AD, Felberg MA, Bidani SA. Validation of the pictorial Baxter Retching Faces scale for the measurement of the severity of postoperative nausea in Spanish-speaking children. Br J Anaesth. 2018 Dec;121(6):1316-1322. doi: 10.1016/j.bja.2018.07.036. Epub 2018 Sep 7. PMID 30442259

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nausea Measurement by VAS and BARF
Started | 193
PACU Analysis | 184
Completed (Post-Discharge Analysis) | 82
Not Completed | 111
Not completed — Diary not returned or excluded | 102
Not completed — Excluded - Age<7yo | 9

BASELINE CHARACTERISTICS:
Arm/Group | Nausea Measurement by VAS and BARF
Number analyzed (Participants) | 184
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 10.9 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74
  Male | 110
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 184
Preoperative VAS Nausea (Normalized Values) [Mean (Full Range); unit: cm] — Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no nausea" and "worst nausea."
  cm | 0.2 [0 to 4.6]
Preoperative VAS Pain (Normalized Values) [Mean (Full Range); unit: cm] — Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."
  cm | 0.4 [0 to 9.3]
Preoperative FACES Pain [Mean (Full Range); unit: units on a scale] — Score the chosen face 0, 2, 4, 6, 8, or 10, counting left to right, so "0" equals "No pain" and "10" equals "Very much pain."
  units on a scale | 0.4 [0 to 6]
Preoperative FACES Nausea [Mean (Full Range); unit: units on a scale] — Score the chosen face 0, 2, 4, 6, 8, or 10, counting left to right, so "0" equals "No nausea" and "10" equals "Very much nausea."
  units on a scale | 0.3 [0 to 4]

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Postoperative Nausea and/or Vomiting (PONV) in the Postanesthesia Care Unit (PACU)
Description: Subjects rated their pain and nausea at these time points: (1) upon waking in the PACU, (2) just before and (3) 30-60 mins after receiving analgesic or antiemetic therapy, and (4) upon discharge from PACU.
  Scales range from 0 to 10 (lower scores indicate no pain or nausea).
Time Frame: When awake and responding to commands in the post-anesthesia care unit (PACU)
Population: Some PACU data is partial due to subjects being uncooperative at times (n=5) or being asleep until just before discharge (n=2)
Measure: Mean (Full Range); unit: units
Groups:
- PACU Time: Subject's rated their pain and nausea while in PACU
- Discharge From PACU: Subjects rated their pain and nausea upon discharge from PACU
Arm/Group | PACU Time | Discharge From PACU
Number analyzed (Participants) | 177 | 175
units
  VAS Nausea | 0.6 [0 to 10] | 0.4 [0 to 7.6]
  VAS Pain | 2.7 [0 to 10] | 1.3 [0 to 9]
  FACES Nausea | 0.9 [0 to 10] | 0.5 [0 to 8]
  FACES Pain | 2.7 [0 to 10] | 1.6 [0 to 10]

2. Secondary Outcome: Subjects Who Experienced Nausea and/or Vomiting After Discharge (PDNV)
Description: The study design is a cross sectional study of patients undergoing surgery. There will be no group assignment, no placebo group and each patient will be his or her own control. All patients will be asked to assess their pain and nausea using the visual analogue scales, the modified faces scale and the BARF scale as described below in the preoperative and postoperative areas.
Time Frame: First 24 postoperative hours
Measure: Count of Participants; unit: Participants
Groups:
- Post-Discharge Analysis: This includes all subjects who returned their diaries.
Arm/Group | Post-Discharge Analysis
Number analyzed (Participants) | 82
Participants | 10

3. Secondary Outcome: Pain and/or Nausea/Vomiting Rescue Needed
Description: Incidence and/of pain or nausea/vomiting rescue medications administered during time in the PACU
Time Frame: Time in the PACU
Measure: Count of Participants; unit: Participants
Arm/Group | Nausea Measurement by VAS and BARF
Number analyzed (Participants) | 184
Participants | 100

ADVERSE EVENTS:
Time Frame: Subjects were monitored for adverse events while active in the study (from enrollment until diaries were completed at 24 hours PACU discharge).
Description: This is a minimal risk, cross-sectional study of pain and nausea using three scales. There was no randomization or intervention.
Arm/Group | Nausea Measurement by VAS and BARF
All-Cause Mortality (participants affected / at risk) | 0/193
Serious Adverse Events (participants affected / at risk) | 0/193
Other Adverse Events (participants affected / at risk) | 0/193

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-07): https://cdn.clinicaltrials.gov/large-docs/09/NCT02007109/Prot_SAP_000.pdf